CLINICAL TRIAL: NCT00747812
Title: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial of Occipital Nerve Stimulation for Drug Refractory Migraine
Brief Title: Study of Occipital Nerve Stimulation for Drug Refractory Migraine
Acronym: PRISM UK
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor closed enrollment early based on interim data from the PRISM US Pivotal Study.
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PRISM-UK-05
Record Dates: First submitted 2008-09-04; First posted 2008-09-05 (Estimated); Results first posted 2012-08-03 (Estimated); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Migraine
Keywords: Headache; Migraine; Refractory; Chronic; Pain
MeSH Terms: conditions — Migraine Disorders; Headache; Bronchiolitis Obliterans Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Stimulation on from activation to 12 weeks post-activation. Stimulation off from 12 weeks post-activation to 16 weeks post-activation. Stimulation on from 16 weeks post-activation to end of study.
  Interventions: Device: Precision
- 2 (Sham Comparator): Sham Stimulation from activation of device to 12 weeks post-activation. Stimulation on from 12 weeks post-activation on.
  Interventions: Device: Precision

INTERVENTIONS:
Device: Precision — Implantable Neurostimulator

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an implantable device to treat migraine. There are a significant number of patients who have drug refractory migraine and alternative therapies are needed.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with multiple migraines per month of moderate to severe intensity;
* Be refractory to medication;
* Be an appropriate candidate for the surgical procedures required fo this study;
* Be willing and able to comply with all study related procedures;
* Be capable of reading and understanding patient information materials and giving written informed consent.

Exclusion Criteria:

* Have onset of headache after age 50;
* Are current substance abusers (including alcohol and illicit drugs);
* Have a significant psychiatric disorder;
* Have previously been treated with occipital nerve stimulation (either temporary trial or permanent implant);
* Have had nerve stimulation for pain relief.
* Have had an injection of botulinum toxin in the head or neck within 6 months prior to enrollment;
* Have previously undergone destructive ganglionectomy affecting C2/C3 occipital and/or trigeminal distribution or have an occipital blockade or radiofrequency procedure currently in effect.
* Have a condition currently requiring or likely to require the use of MRI or diathermy;
* Have an active implantable device;
* Are pregnant or lactating or planning to become pregnant in the next 14 months;
* Have participated in any drug or device trial in the last 4 weeks or plant to participate in any other study during the next 14 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-05; Primary Completion 2008-11 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter J. Goadsby, MD, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital - Dept of Clinical Neurosciences, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Active Stimulation (Treatment Group): Stimulation on from activation to 12 weeks post-activation. Stimulation off from 12 weeks post-activation to 16 weeks post-activation. Stimulation on from 16 weeks post-activation to end of study.
- Sham Stimulation (Control Group): Sham Stimulation from activation of device to 12 weeks post-activation. Stimulation on from 12 weeks post-activation on.
Period: Overall Study
Arm/Group | Active Stimulation (Treatment Group) | Sham Stimulation (Control Group)
Started | 5 | 3 (4 subjects were randomized to the Control Group; 1 was not implanted due to early enrollment closure)
Completed | 0 | 0
Not Completed | 5 | 3
Not completed — Research Site Staff Relocation | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation (Treatment Group) | Sham Stimulation (Control Group) | Total
Number analyzed (Participants) | 5 | 3 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (15.5) | 55.6 (5.5) | 50.7 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 6
  Male | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United Kingdom | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Hours of Headache
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: Hours
Groups:
- Active Stimulation (Treatment Group): Active stimulation from IPG activation to 12 weeks post-IPG activation. Stimulation off from 12 weeks post-activation to 16 weeks post-activation. Stimulation on from 16 weeks post-activation to end of study.
- Sham Stimulation (Control Group): Sham stimulation from IPG activation to 12 weeks post-IPG activation. Stimulation on from 12 weeks post-activation on.
Arm/Group | Active Stimulation (Treatment Group) | Sham Stimulation (Control Group)
Number analyzed (Participants) | 5 | 3
Hours | NA (NA) — Efficacy endpoint data for this study was not analyzed because of the amount of insufficient data collected from the limited number of implanted subjects. | NA (NA) — Efficacy endpoint data for this study was not analyzed because of the amount of insufficient data collected from the limited number of implanted subjects.

2. Primary Outcome: Number of Days With 4 or More Hours of Headache
Time Frame: 12 Weeks
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Active Stimulation (Treatment Group) | Sham Stimulation (Control Group)
Number analyzed (Participants) | 5 | 3
Days | NA (NA) — Efficacy endpoint data for this study was not analyzed because of the amount of insufficient data collected from the limited number of implanted subjects. | NA (NA) — Efficacy endpoint data for this study was not analyzed because of the amount of insufficient data collected from the limited number of implanted subjects.

ADVERSE EVENTS:
Arm/Group | Active Stimulation (Treatment Group) | Sham Stimulation (Control Group)
Serious Adverse Events (participants affected / at risk) | 4/5 | 2/4
Other Adverse Events (participants affected / at risk) | 5/5 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (Treatment Group) (N=5) | Sham Stimulation (Control Group) (N=4)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Joint Range of Motion Decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Therapeutic Product Ineffective (General disorders) | 2 (2) | 0 (0)
Implant Site Pain (General disorders) | 1 (1) | 0 (0)
Umbilical Hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Device Ineffective (General disorders) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (Treatment Group) (N=5) | Sham Stimulation (Control Group) (N=4)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Impaired healing (General disorders) | 1 (1) | 0 (0)
Implant site pain (General disorders) | 1 (1) | 0 (0)
Implant site reaction (General disorders) | 2 (2) | 1 (1)
Inflammation (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0)
Incision site infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Device failure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Gastrointestinal disorder postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Inappropriate device stimulation of tissue (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Incision site complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Incision site pain (Injury, poisoning and procedural complications) | 4 (4) | 1 (1)
Medical device pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Wound secretion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Dysaesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Head discomfort (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2)
Syncope vasovagal (Nervous system disorders) | 1 (1) | 0 (0)
Sleep disorder (Psychiatric disorders) | 2 (2) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Nail disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Onychalgia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Insufficient data collected from limited number of implanted subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No